CLINICAL TRIAL: NCT05217628
Title: A Phase II/III, Multicentre, 8-week run-in Phase Followed by a 12-week, Prospective, Parallel-group, Double-blind, Randomized Withdrawal, Placebo-controlled Study, With a 52 Week Open Label Extension, to Evaluate the Efficacy and Safety of Daily 1.5 to 3.5 mg Basimglurant in Patients With Pain Associated With Trigeminal Neuralgia With Suboptimal Response to Their Current Anti-pain Therapy.
Brief Title: An Efficacy and Safety Study of Basimglurant (NOE-101) in Patients With Trigeminal Neuralgia.
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Noema Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NOE-TGN-201
Record Dates: First submitted 2021-12-15; First posted 2022-02-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Trigeminal Neuralgia
MeSH Terms: conditions — Trigeminal Neuralgia | interventions — 2-chloro-4-(1-(4-fluorophenyl)-2,5-dimethyl-1H-imidazol-4-ylethynyl)pyridine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Basimglurant/NOE-101 (Experimental): * Period 1 (Run-in: Baseline1 to Week 8): Basimglurant once daily dosing starting dose 1.5mg
  * Period 2 (Double blind: Weeks 9 to 20): Participants will receive double-blind treatment with Basimglurant once daily.
  * Open-label Extension (OLE): On completion of Period 2, participants will be offered open label treatment with Basimglurant in an open label extension for up to 52 weeks.
  Interventions: Drug: Basimglurant
- Arm B: Placebo (Placebo Comparator): - Period 2 (Double blind: Week 9 to Week 20): Participant randomized to placebo will receive the corresponding number of matching placebo capsules.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Basimglurant — Period 1: Basimglurant 1.5 to 3.5 mg QD titrated on individual tolerability.
  Period 2: Patients randomized to receive either double blind Basimglurant at the tolerated dose from Period 1 or Placebo.
  OLE: Open label Basimglurant at the dose tolerated from Period 2, patients previously assigned placebo in period to be titrated to the Period 1.
  Other Names: NOE-101
  Arms: Arm A: Basimglurant/NOE-101
Other: Placebo — Participant randomized to receive matching placebo once daily.
  Arms: Arm B: Placebo

SUMMARY:
Trigeminal neuralgia (TN), also called "tic douloureux", is the most common form of craniofacial neuropathic pain and is considered the cause of one of the most painful afflictions known in medical practice.

This study is designed to evaluate the efficacy and safety of 1.5mg - 3.5mg basimglurant in adults with TN.

DETAILED DESCRIPTION:
This study is designed to evaluate the efficacy and safety of basimglurant (NOE-101) in patients with TN. Basimglurant is a potent inhibitor of metabotropic glutamate receptor 5 (mGluR5) which controls a wide range of processes in both central and peripheral nervous system. Inhibition of the mGluR5 receptor has shown therapeutic potential for pain associated with conditions such as TN. The drug has been shown to have a favorable safety profile in adults, children and adolescents. The aim of the study is to determine whether Basimglurant decreases both duration and intensity of facial pain associated with TN by use of a patient pain diary and the Patient-reported Global Impression of Change (PGI-C) compared to baseline.

ELIGIBILITY:
Inclusion Criteria (Summary):

1. Ability and willingness to provide written informed consent and to comply with the study procedures.
2. Fluency in the language of the investigator, study staff and the informed consent.
3. Age 18-75 years.
4. Diagnosis of primary trigeminal neuralgia (TN) as per the ICHD-3 criteria confirmed by the study neurologist.
5. Experience pain due to TN and at baseline, experience at least 3 paroxysms per day of at least intensity of 4 or more on a pain intensity numerical rating scale (PI-NRS) during the last 7 days.
6. Female patients who are either sterile or menopausal. For female patients with childbearing potential, must be neither pregnant nor lactating (with appropriate contraceptive precautions and prior negative pregnancy tests).

Exclusion Criteria (Summary):

Patients who meet any of the following criteria will be excluded from participation in this study:

1. Current or prior history of any major psychiatric diagnoses unrelated to TN. Patients with TN-related depressive symptoms are permitted.
2. Current or prior history of mania, or psychotic episodes.
3. History of DSM-5-defined substance dependence and/or substance abuse in the last six months [180 days], except for nicotine.
4. Patient not willing to discontinue their current TN analgesic medication.
5. Use of opioids, except for pain control on a prn basis as long as it does not exceed 2 days per week.
6. Known allergic reaction to the investigational drug or one of its components.
7. Patients with secondary TN as per the ICHD-3 criteria.

   Medication history:
8. Previous treatment with basimglurant, except with the prior agreement of the medical monitor.
9. Treatment with antipsychotics within six months (180 days) of screening.
10. Any investigational drug within 90 days prior to initiation of study drug.

    Medical status:
11. Evidence of clinically significant, uncontrolled, unstable medical conditions or recently diagnosed cardiovascular disease, such as ischemic heart disease, coronary artery vasospasm, and cerebral ischemia. Subjects with myocardial infarction, acute coronary syndrome, percutaneous coronary intervention, cardiac surgery, stroke or transient ischemic attack during the 6 months prior to screening.
12. Subject has a history of gastric, or small intestinal surgery (including gastric bypass, gastric banding, gastric sleeve, gastric balloon, etc.) that may, in the opinion of the investigator, may cause malabsorption, or has a disease of the GI tract that causes malabsorption.
13. Body mass index > 39kg/m²
14. Patients with moderate or severely impaired hepatic function, ie, Pugh-Child score C.
15. Patients with severe renal impairment, ie, eGFR or creatinine clearance lower than 30mL/min.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2022-01-11 (Actual); Primary Completion 2027-02-02 (Estimated); Study Completion 2027-04-24 (Estimated)

PRIMARY OUTCOMES:
Period 1: Incidence and severity of adverse events, laboratory, vital signs and cardiovascular events. | 8 weeks
  Change in pain as measured by the pain diary (TnED).
Period 2: Time to Loss of Efficacy or pain recurrence defined as the confirmed increase in the number of weekly paroxysms or re-emergence of continuous pain and/or the need for rescue medication. | 12 weeks
  To assess the maintenance of effect on pain.
Open Label Extension: Incidence and severity of adverse events, laboratory, vital signs and cardiovascular events. | 52 weeks
  To evaluate the long-term safety of basimglurant daily dosing.

SECONDARY OUTCOMES:
Period 2: Mean change in the total patient-rated Penn-Facial Pain Scale-Revised (Penn-FPS-R) scale compared with Period 2 baseline (BL2). | 12 weeks
  Impact on facial pain.
Period 2: Frequency of attacks (paroxysms). | 12 weeks
  Impact on facial pain measured by patient rated scale via Penn-FPS-R
Period 2: Severity of attacks (paroxysms). | 12 weeks
  Impact on facial pain measured by patient rated scale via Penn-FPS-R
Period 2: Severity of continuous pain. | 12 weeks
  Impact on facial pain measured by patient rated scale via Penn-FPS-R
Period 2: Duration of continuous pain. | 12 weeks
  Impact on facial pain measured by patient rated scale via Penn-FPS-R
Period 2: Change in Patient Global Impression of Change (P-GIC). | 12 weeks
  Impact on facial pain.
Period 2: Change in Medication Satisfaction Questionnaire (MSQ). | 12 weeks
  Impact on facial pain.
Open Label Extension: Frequency of attacks (paroxysms). | 52 weeks
  Evaluate the continued efficacy of basimglurant on facial pain measured by patient rated scale via Penn-FPS-R
Open Label Extension: Severity of attacks (paroxysms). | 52 weeks
  Evaluate the continued efficacy of basimglurant on facial pain measured by patient rated scale via Penn-FPS-R
Open Label Extension: Severity and duration of continuous pain reported in patient pain diary. | 52 weeks
  Evaluate the continued efficacy of basimglurant on facial pain.
Open Label Extension: Measure Global Impression of Severity as captured by PGI-S. | 52 weeks
  Evaluate the continued efficacy of basimglurant on facial pain.

OTHER OUTCOMES:
Period 1: Mean change from Period 1 baseline (BL1) to Week 8 in the total patient-rated Penn-Facial Pain Scale-Revised (Penn-FPS-R) scale. | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Measure Global Impression of change from Period 1 baseline (BL1) to Week 8. | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Number and severity of attacks (paroxysms). | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Duration of continuous pain compared with BL1. | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following as measured by patient rated scale via Penn-FPS-R:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Severity of continuous pain compared with BL1. | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following as measured by patient rated scale via Penn-FPS-R:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Number of pain free days. | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 1: Patient reported rating of the Medication Satisfaction Questionnaire (MSQ). | 8 weeks
  Evaluate 8-week once daily basimglurant on pain associated with TN on the following:
  * Impact on Facial Pain
  * Patient perceived change of the pain
  * Pain assessments
  * Pain freedom
  * Patient medication satisfaction
Period 2: The impact of pain on general activities of daily living captured in patient diary cards. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (34):
- United States (8):
  - Kaizen Brain Center (Site #: 1001), La Jolla, California
  - L & A Morales Healthcare INC (Site#: 1011), Miami, Florida
  - University of South Florida (Site #: 1002), Tampa, Florida
  - Vista Clinical Research,LLC (Site#: 1010), Newnan, Georgia
  - Beth Israel Deaconess Medical Center (Site #: 1004), Boston, Massachusetts
  - Altea Research - Nevada - ClinEdge - PPDS (Site #1006), Las Vegas, Nevada
  - Columbia University - Irving Medical Center (Site #: 1008), New York, New York
  - University of Cincinnati (Site #: 1007), Cincinnati, Ohio
- Danish Headache Center (Site #: 1201), Glostrup Municipality, Denmark
- Universitätsklinikum Bonn (Site #: 1707), Bonn, Germany
- Italy (5):
  - Università Campus Bio Medico Di Roma (Site #: 1805), Rome, Lazio
  - IRCCS San Raffaele Pisana (Site #: 1801), Rome, Lazio
  - La Sapienza-Università di Roma-Policlinico Umberto I (Site #: 1802), Rome, Lazio
  - Azienda Ospedaliera Universitaria Careggi (Site #: 1806), Florence
  - Fondazione IRCCS Di Rilievo Nazionale Istituto Nazionale Neurologico Carlo Besta (Site #: 1804), Milan
- Poland (5):
  - Niepubliczny Zaklad Opieki Zdrowotnej (NZOZ) Zespo (Site #: 2602), Dąbrowa Górnicza
  - Centrum Medyczne Linden (Site #: 2605), Krakow
  - FutureMeds - Lodzi - PPDS (Site #: 2606), Lodz
  - Prywatny Gabinet Lekarski U. Chyrchel-Paszkiewicz (Site #: 2604), Lublin
  - MIGRE Polskie Centrum Leczenia Migreny Anna Gryglas-Dworak (Site #: 2601), Wroclaw
- Spain (4):
  - Hospital Universitario Fundacion Jimenez Diaz (Site #: 1903), Madrid, Madrid
  - Hospital Universitario La Paz - PPDS (Site #: 1907), Madrid, Madrid
  - Hospital Universitario Virgen del Rocio - PPDS (Site #: 1904), Seville, Sevilla
  - Hospital Clinico Universitario de Valencia (Site #: 1906), Valencia, Valencia
- Turkey (Türkiye) (8):
  - Duzce University Health Application and Research Center (9008), Düzce, Düzce
  - Selcuk University Medical Faculty (Site #: 9006), Selçuklu, Konya
  - Afyon Kocatepe University Faculty of Medicine (Site #: 9005), Afyonkarahisar
  - Uludag University Faculty of Medicine Hospital (Site #: 9001), Bursa
  - Istanbul University Istanbul Medical Faculty Hospital (Site #: 9003), Istanbul
  - Bagcilar Medipol Mega University Hospital (Site #: 9002), Istanbul
  - Kocaeli University Faculty of Medicine Hospital (Site #: 9004), Kocaeli
  - Mersin University Faculty of Medicine Hospital (Site #: 9007), Mersin
- United Kingdom (2):
  - St. Thomas' Hospital (Site #: 2504), London, London
  - St Pancras Clinical Research (Site #: 2503), London, Middlesex